CLINICAL TRIAL: NCT06356935
Title: Effects of Resistance Training on Lower Limb Mechanical Muscle Function and Sports Specific Performance in Elite Female Team Handball Players
Brief Title: Effects of Heavy-load Resistance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Team Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP2024
Record Dates: First submitted 2024-03-26; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: Resistance training; Agility performance; Jump capacity; Knee extensor and flexor strength; Explosive muscle strength; Sprint ability

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance training (Experimental): Assigned to heavy-load undulating resistance training.
  Interventions: Other: RT
- Control (Active Comparator): Training-as-usual off-season strength and conditioning training, programs provided by respective clubs
  Interventions: Other: CON

INTERVENTIONS:
Other: RT — Resistance training
  Arms: Resistance training
Other: CON — Control group
  Arms: Control

SUMMARY:
The study aims to investigate effects of 8-weeks of heavy-load resistance training on mechanical muscle function and functional performance in elite female team handball players from the Danish Women's Handball League. Players will be randomly assigned to either a resistance training group (RT) or serves as training-as-usual controls (CON).

DETAILED DESCRIPTION:
The study aims to examine how an eight-week heavy-load resistance training regimen affects both mechanical muscle function and functional performance in elite female team handball players. Given the sport's demands for rapid and forceful muscle actions, understanding the impact of such training on functional performance is crucial.

Players from four clubs in the Danish Women's Handball League, will be randomly block randomized (one block=one club) into two groups: the heavy-load resistance training group (RT), and the control group (CON). Each group contains players from 2 clubs. The study will conduct a battery of tests to evaluate various aspects of mechanical muscle function and performance, including isometric knee extensor and flexor peak torque, countermovement jump (CMJ) power/work, and functional measures like sprinting, jump height, and agility performance.

ELIGIBILITY:
Inclusion Criteria:

* Playing in the Danish Women's Handball League.

Exclusion Criteria:

* Absent from team handball training for more than two weeks due to injuries, within the six months preceding PRE-testing.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-17 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Explosive muscle strength | Eight week off-season
  Rate of torque development - (Nm/s)/kg
Acceleration capacity | Eight week off-season
  Sprint performance - seconds
Agility performance | Eight week off-season
  Game-based agility performance - seconds
Jump ability | Eight week off-season
  Countermovement jump height - cm

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Fristrup, MSc, Principal Investigator — Department of Sports Science and Clinical Biomechanics, University of Southern Denmark
Locations (1):
- University of Southern Denmark, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No